CLINICAL TRIAL: NCT01241487
Title: An 8 Weeks Open Label National Multicentre Study to Assess the Efficacy of the Fixed Combination of Valsartan and Amlodipine in Hypertensive Patients Not Controlled by Monotherapy
Brief Title: A National Multicentre Study to Assess the Efficacy of the Fixed Combination of Valsartan and Amlodipine in Hypertensive Patients Not Controlled by Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489AEG02
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Primary Hypertension
Keywords: Hypertension, Valsartan/Amlodipine,
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): valsartan/amlodipine
  Interventions: Drug: valsartan/amlodipine

INTERVENTIONS:
Drug: valsartan/amlodipine — 160/10 mg

SUMMARY:
This study is to assess the efficacy of the fixed combination of Valsartan and Amlodipine in hypertensive patients uncontrolled by monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient uncontrolled by mono-therapy for at least 8 weeks, having B.P.>/= 140/90 mmHg in non diabetics or >/= 130/80 mmHg in diabetics

Exclusion Criteria:

* Patient having B.P.>= 180/110 mmHg in non diabetics or >= 160/100 mmHg in diabetics
* Type 1 Diabetes or uncontrolled type 2 Diabetes.
* PCI in last 12 months.
* Concomitant unstable angina. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Hypertension in patients that will be controlled on each concentration and those that will switch to the higher concentration (160/10) | 4 weeks

SECONDARY OUTCOMES:
Hypertension of patients that were previously controlled on (160/5) and those that were uncontrolled and switched to the higher concentration (160/10) after 4 weeks on (160/5) concentration. | 8 weeks
Safety and Tolerability of the Trial Medication | 8 weeks
The incidence of Edema | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Dr Ahmed Anwar Clinic,, Cairo, Egypt